CLINICAL TRIAL: NCT03883347
Title: Sedation With Dexmedetomidine Versus Remifentanil in Urogynecological Surgery Under Spinal Anaesthesia : Impact on Block Characteristics, on Acute and Chronic Postoperative Pain
Brief Title: Sedation With Dexmedetomidine Versus Remifentanil in Urogynecological Surgery Under Spinal Anaesthesia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Staikou Chryssoula, Assistant Professor of Anesthesiology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 107/13-02-2019
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Vaginal Hysterectomy; Suburethral Slings
MeSH Terms: interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All syringes and solutions will be prepared by an independent researcher who will not be further involved in the study eg data collecting or analyzing them.All syringes will look identical to the anesthetist who will administer them to the patients.Apart from the anesthetist, the surgery staff and the researchers recording the measurements will not know the therapeutic intervention team in which each patient has been randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DEX (Active Comparator): Intravenous administration of dexmedetomidine 0.6 mcg / kg within 10 minutes prior to regional anesthesia. The infusion of the solution will be discontinued and then will be performed in all patients subarachnoid anesthesia. Starting with Tmax, infusion of the solution will be initiated again at a dose of 0.6 mcg / kg / h.
  Interventions: Drug: Dexmedetomidine
- Group REMI (Active Comparator): Intravenous administration of remifentanil 1 mcg / kg within 10 minutes prior to regional anesthesia. The infusion of the solution will be discontinued and then will be performed in all patients subarachnoid anesthesia. Starting with Tmax, infusion of the solution will be initiated again at a dose of 0.025 mcg / kg / min.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Intravenous administration of dexmedetomidine 0.6 mcg / kg within 10 minutes prior to regional anesthesia and 0.6 mcg / kg / h after performing regional anaesthesia until the end of the surgery
  Other Names: DEXDOR
  Arms: Group DEX
Drug: Remifentanil — Intravenous administration of remifentanil 1 mcg / kg within 10 minutes prior to regional anesthesia and 0.025 mcg / kg / h after performing regional anaesthesia until the end of the surgery
  Other Names: ULTIVA
  Arms: Group REMI

SUMMARY:
Neuraxial blocks are usually used as an anaesthetic method for urogynecological surgeries. In most patients under regional anaesthesia, premedication is given for reducing anxiety. Purpose of this prospective double blind randomised clinical trial is the investigation of the effect of perioperative intravenous infusion of dexmedetomidine vs remifentanil for sedation in patients under spinal anaesthesia for urogynecological procedures.

DETAILED DESCRIPTION:
The day before surgery the procedure will be explained to the patient and the written consent will be obtained. In the operating room, intraoperative monitoring will include ECG, noninvasive blood pressure, oxygen saturation by pulse oximetry (SpO2) and heart rate (HR). A peripheral intravenous catheter wil be placed for fluid replacement ( Ringer's Lactate solution 6 - 8ml/ kg/hr) and administration of drugs.

Women will be randomly assigned into one of two groups:

Group A: Women will receive dexmedetomidine continuously infused at a dose of 0,6 mcg/kg for 10 minutes (concentration of the solution 6mcg/ml) before spinal anaesthesia. Infusion will be stopped in order to proceed with regional anesthesia.

Group B: Women will receive remifentanil continuously infused at a dose of 1mcg/kg for 10 minutes (concentration of the solution 1mcg/ml) before spinal anaesthesia. Infusion will be stopped in order to proceed with regional anesthesia.

The insertion of a 27 Gauge (27G) spinal needle is performed at L3-L4 or L4-L5 interspace, in the lateral position. All patients will receive 2,7 ml ropivacaine 0,75% and 15 mcg fentanyl intrathecally and assessment of sensory and motor block will be assessed every 2 min. The moment that sensory block is in the highest dermatome and motor block is complete (Bromage grade 3) is Time to max effect (Tmax). In group A an infusion of dexmedetomidine (6mcg/ml) at a dose of 0,6mcg/kg/hr will be administered and in group B an infusion of remifentanil (1mcg/ml) at a dose of 0,03 mcg/kg/min.At the end of the surgery patients will be transferred in Post Anaesthetic Care Unit (PACU) and a patient control analgesia (PCA) pump will be provided to the patient, administering 1 mg of morphine in every attempt, with a lock out interval of 10 minutes.There will be no continuous infusion. All patients will receive a standardized multimodal approach, including diclofenac 50 mg t.i.d, paracetamol 1gr as rescue analgesia (max 4 gr per day) and PCA with morphine.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-II
* Patients scheduled for transvaginal urogynecological or gynecological surgery

Exclusion Criteria:

* Patient refusal
* Contraindication of spinal anaesthesia (Coagulopathy, Local infection at the site of injection, Local anaesthetic allergy, Hypovolaemia)
* BMI > 30 kg/m2
* Personal history of cardiovascular disease
* Arrythmias
* Conduction disorders
* Severe kidney or liver dysfunction
* Insulin-dependent diabetes mellitus
* Central nervous system disorders
* Psychiatric and mental status disorders
* Chronic Excessive Alcohol Consumption
* Chronic Use of Opioid Analgesics
* Chronic Use of corticosteroids
* Chronic Use of clonidine (or other a2 adrenergic agonist)
* Use of drugs acting on central nervous system or analgetics the last two weeks
* Communication problems due to language barriers or unable to understand the pain scale

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 24 hours postoperatively
  Time for first analgesia / PCA first bolus

SECONDARY OUTCOMES:
Analgesic consumption | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Morphine consumption in mg

OTHER OUTCOMES:
Postoperative pain | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Numerical Rating Scale (NRS scale) (0:no pain 10:worst pain ever)
Chronic pain | 6 months
  Using of Graded Chronic Pain Scale (GCPS) Grade 0: No pain in prior 6 months Grade 1: Low Intensity - Low Disability Grade II: High Intensity Characteristic Pain Intensity - Low Disability Grade III: High Disability - Moderately Limiting Grade IV: High Disability - Severely Limiting
Adverse effects | 24 hours postoperatively
  Adverse effects of drugs, anaesthetic or surgical technique and any intraoperative adverse events
Sedation | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Ramsay sedation scale ( 1:anxious, agitated or restless- 6: asleep, no response )
Postoperative need of rescue analgesia | 24 hours postoperatively
  Consumption of paracetamol
Patient satisfaction over anaesthesia | 24 hours postoperatively
  scale for satisfaction (0:no satisfaction at all, 10:satisfaction)
Nausea | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Scale for nausea (0:no nausea 10:worst possible nausea)
Vomiting | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Number of vomits
Sedation | Baseline (before start of infusion), at 5 minutes load, end of 10 minutes load, at spinal time, every 5 minutes until 30 minutes, every 10 minutes until the end of the surgery
  Ramsay sedation scale(1:anxious, agitated or restless- 6: asleep, no response)
Sensory blockade | 30 minutes
  Time for onset of sensory block at T10 and to maximum sensory block
Motor blockade | 30 minutes
  Time to bromage 2 and to bromage 3
Highest level of sensory block | 30 minutes
  dermatome
Sensory Regression | 240 minutes
  Time to two segment regression
Motor block regression | 240 minutes
  time to bromage 1 and bromage 0
Time to max effect (Tmax) | 30 minutes
  Time when the motor blockade is complete and sensory blockade is in the highest dermatome

CONTACTS AND LOCATIONS:
Overall Officials: Cryssoula Staikou, Principal Investigator — Aretaieio Hospital Medical School University of Athens
Locations (1):
- Aretaieio Hospital, University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No